CLINICAL TRIAL: NCT02393313
Title: Examination of Rayner T-flex Toric Intra-Ocular Lens for Spherical and Astigmatic Correction, and Rotational Stability
Brief Title: Rayner Toric IOL Rotational Stability
Acronym: Rayner-toric
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Rayner Intraocular Lenses Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0670-14-TLV
Record Dates: First submitted 2014-12-08; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Cataract; Corneal Astigmatism
MeSH Terms: conditions — Cataract; Astigmatism | interventions — Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cataract surgery toric intraocular lens (Experimental): Rayner T-flex Toric IOLs (573T / 623T; Rayner Intraocular Lenses Ltd,East Sussex, United Kingdom) will be implanted in the lens capsule
  Interventions: Procedure: Cataract surgery; Device: Rayner T-flex Toric IOLs

INTERVENTIONS:
Procedure: Cataract surgery — Rayner T-flex Toric IOLs (573T / 623T; Rayner Intraocular Lenses Ltd,East Sussex, United Kingdom) will be implanted in the lens capsule
Device: Rayner T-flex Toric IOLs

SUMMARY:
This study evaluates the Rayner T-flex Toric IOLs for spherical and astigmatic correction, and rotational stability in cataract surgery. 50 patients with cataract and corneal astigmatism >= 2 diopters will undergo cataract surgery, with implantation of Rayner toric intraocular lens. Post-operative examination will include IOL axis measurements and refraction.

DETAILED DESCRIPTION:
Background During cataract surgery, an intraocular lens is implanted in the bag. A monofocal lens allows spherical correction only. 15% to 29% of patients with cataracts have more than 1.50 diopters of astigmatism according to current estimations.1 Astigmatic correction can be performed during cataract surgery: the main clear corneal incision can be done at the steep axis, limbal relaxing incisions (LRI) or by opposite clear corneal incision (OCCI) can be performed. These techniques are not fully predictable and stable over time.2 Optimal corneal astigmatic correction can be done by implantation of a toric intra-ocular lens(IOL), with predictable and stable results over time. The toric IOL must be positioned in the correct axis. Rotation of the lens will reduce the astigmatic correction. Approximately one degree of off-axis rotation results in a loss of up to 3.3% of the cylinder power. 3 It is crucial for the intraocular lens to keep its correct axis for optimal astigmatic correction.

A number of toric intraocular lens are approved for implantation such as - Acrysof toric (Alcon), Tecnis toric IOL (Abbott medical), STAAR toric IOL (STAAR surgical company). This study will examine T-flex (Rayner) IOL. The rotational and refractive stability of this IOL has been tested on a relatively small number of patients. 4, 5

Objective Examination of Rayner T-flex Toric IOLs (573T and 623T; Rayner Intraocular Lenses Ltd,East Sussex, United Kingdom) for spherical and astigmatic correction, and rotational stability.

Methods Prospective study on 50 eyes. Patients will be recruited during examination in pre-operative clinic. This examinations include visual acuity, slit-lamp biomicroscopy, applanation tonometry, fundus examination after instillation of tropicamide 0.5% and phenylephrine 10%, IOL calculation with IOLMaster(Zeiss), which also measures corneal astigmatism. After acquiring informed consent, further examinations will be done including corneal topography with Galilei Dual Scheimpflug Analyzer ( Zeimer Ophthalmology), and Tomey keratometer, auto-refractometry and subjective refraction.

Since corneal astigmatism is often binocular, patients with second eye corneal astigmatism, will be offered a toric IOL, even if unsuitable for inclusion in this study. All operations will be done by a senior surgeon, experienced in toric IOL implantations. Rayner T-flex Toric IOLs (573T / 623T; Rayner Intraocular Lenses Ltd,East Sussex, United Kingdom) will be implanted. IOL calculation will be done using Ranyer's online calculator (WWW.TORICIOL.RAYNER.COM).

Post-operative examination will include IOL axis measurements, IOL photography and refraction after a week, month and three months.

ELIGIBILITY:
Inclusion Criteria:

* Corneal astigmatism ≥ 2.00 measured by IOLMaster

Exclusion Criteria:

* Pterygium (can be included 6 months after successful surgical excision)
* Corneal pathologies including corneal scars causing corneal irregularity
* Severe dry eye
* Traumatic cataract
* Pregnant women
* Severe macular disease or macular atrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
IOL off-axis rotation | 3 months after surgery
  IOL axis will be measured by slit lamp biomicroscopy and compared to the planned axis

SECONDARY OUTCOMES:
Uncorrected distance visual acuity | 3 months after surgery
Corrected distance visual acuity | 3 months after surgery
Subjective refraction | 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Adi Michaeli, MD, Principal Investigator — michaeli.adi@gmail.com
Locations (1):
- Departent of Ophthalmlogy, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Background] Hoffer KJ. Biometry of 7,500 cataractous eyes. Am J Ophthalmol. 1980 Sep;90(3):360-8. doi: 10.1016/s0002-9394(14)74917-7. No abstract available. PMID 7425052
- [Background] Tehrani M, Dick HB. Incisional keratotomy to toric intraocular lenses: an overview of the correction of astigmatism in cataract and refractive surgery. Int Ophthalmol Clin. 2003 Summer;43(3):43-52. doi: 10.1097/00004397-200343030-00005. No abstract available. PMID 12881648
- [Background] Becker KA, Auffarth GU, Volcker HE. [Measurement method for the determination of rotation and decentration of intraocular lenses]. Ophthalmologe. 2004 Jun;101(6):600-3. doi: 10.1007/s00347-003-0951-7. German. PMID 15197576
- [Background] Entabi M, Harman F, Lee N, Bloom PA. Injectable 1-piece hydrophilic acrylic toric intraocular lens for cataract surgery: efficacy and stability. J Cataract Refract Surg. 2011 Feb;37(2):235-40. doi: 10.1016/j.jcrs.2010.08.040. PMID 21241904
- [Background] Alberdi T, Macias-Murelaga B, Bascaran L, Goni N, de Arregui SS, Mendicute J. Rotational stability and visual quality in eyes with Rayner toric intraocular lens implantation. J Refract Surg. 2012 Oct;28(10):696-701. doi: 10.3928/1081597X-20120921-04. PMID 23061999